CLINICAL TRIAL: NCT01713985
Title: Feasibility Study: Evaluation of the Ulthera® System vs Thermage® for Lifting and Tightening of the Full Face and Neck
Brief Title: Feasibility Study: Evaluation of Ulthera Versus Thermage for Treating the Face and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-135
Record Dates: First submitted 2012-10-15; First posted 2012-10-25 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-09

CONDITIONS: Skin Laxity; Wrinkles
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Ulthera System Treatment Right, Thermage Left
  Interventions: Device: Ulthera System Treatment; Device: Thermage
- Group B (Active Comparator): Ulthera System Treatment Left, Thermage Right
  Interventions: Device: Ulthera System Treatment; Device: Thermage

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™
Device: Thermage — Radiofrequency treatment focusing radiofrequency energy

SUMMARY:
Up to 20 subjects will be enrolled and randomly assigned to one of two treatment groups. Group A will receive Ultherapy™ on the right side of the face and neck and Thermage on the left side. Group B will receive Thermage on the right side of the face and neck and Ultherapy™ on the left side. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, double-blinded, split-face, randomized pilot study. A triple Ultherapy® treatment and standard Thermage treatment will be provided to all subjects to the full half face, neck, and submental areas. Changes in face and neck skin laxity and wrinkles, from baseline and between study treatments, will be assessed at study follow-up visits. Patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years.
* Subject in good health.
* Skin laxity on the area(s) to be treated.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the area(s) to be treated.
* Excessive skin laxity on the area(s) to be treated.
* Significant scarring in the area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Presence of a metal stent or implant in the area(s) to be treated.
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within two weeks prior to study participation or during the study.
* Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* BMI equal to or greater than 25.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Lifting and Tightening of Skin | 180 days post treatment
  Determined by a masked, qualitative assessment of photographs at 180-days post-treatment compared to baseline. Improvement in skin laxity will be assessed based on photographs taken using the 3D Vectra digital imaging system.
Number of Participants with Wrinkle Reduction | 180 days post treatment
  Determined by a masked, qualitative assessment of photographs at 180-days post-treatment compared to baseline. Improvement in wrinkle reduction will be assessed based on photographs taken using the 3D Vectra digital imaging system

SECONDARY OUTCOMES:
Number of Participants with Eyebrow Lift | 90 days post-treatment
  Quantitative measurements of eyebrow lift will be obtained at follow-up compared to baseline.
Number of Participants with Lower face and Neck Lift | 90 days post-treatment
  Quantitative measurements of lower face and neck lift will be obtained at follow-up compared to baseline.
Number of Participants Reporting Treatment Satisfaction | 180 days post-treatment
  Subjects will complete a split-face Patient Satisfaction Questionnaire at 180 days following study treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Faces+
Locations (1):
- FACES+, San Diego, California, United States